CLINICAL TRIAL: NCT04756193
Title: Evaluate Long Term Cardiovascular and Pulmonary Complications After COVID-19 With Point of Care Ultrasound
Status: Completed | Type: Observational
Sponsor: University of Louisville (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Jiapeng Huang, Professor, MD, PhD, University of Louisville
Other Study IDs: 20.0836
Record Dates: First submitted 2021-02-07; First posted 2021-02-16 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Covid19; Echocardiography; Ultrasound
MeSH Terms: conditions — COVID-19 | interventions — Electrocardiography; Oximetry; Blood Specimen Collection; Spirometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Asymptomatic/Mild COVID-19 Group: 50 confirmed COVID-19 patients who showed no or only mild respiratory/GI symptoms (not admitted to the hospital at all)
  Interventions: Diagnostic Test: Point of care ultrasound including echocardiography, lung ultrasound, vascular ultrasound
- Moderate COVID-19 Group: 50 confirmed COVID-19 patients who were able to maintain oxygen saturation above 92% (or above 90% for patients with chronic lung disease) with up to 4 L/min oxygen via nasal prongs (admitted to the hospital, but never to the ICU and no obvious cardiac complications during the stay)
  Interventions: Diagnostic Test: Point of care ultrasound including echocardiography, lung ultrasound, vascular ultrasound
- Severe COVID-19 Group: 50 confirmed COVID-19 patients who had oxygen saturation lower than 92% at rest and PaO2/FiO2 between 200 and 300 (High-flow oxygen group, mostly in the ICU, and may have some cardiac complications)
  Interventions: Diagnostic Test: Point of care ultrasound including echocardiography, lung ultrasound, vascular ultrasound
- Critical COVID-19 Group: 50 confirmed COVID-19 patients who had PaO2/FiO2 less than 200 or required mechanical ventilation (in the ICU, need mechanical ventilation and more likely to have cardiac complications)
  Interventions: Diagnostic Test: Point of care ultrasound including echocardiography, lung ultrasound, vascular ultrasound
- Control Group: 50 age and sex-matched controls from our hospital admission database
  Interventions: Diagnostic Test: Point of care ultrasound including echocardiography, lung ultrasound, vascular ultrasound

INTERVENTIONS:
Diagnostic Test: Point of care ultrasound including echocardiography, lung ultrasound, vascular ultrasound — Point of care ultrasound including echocardiography, lung ultrasound, vascular ultrasound, ECG, pulse oximetry, blood draw, spirometry
  Other Names: ECG, pulse oximetry, blood draw, spirometry

SUMMARY:
We hypothesize that recovered COVID-19 patients suffer long term cardiovascular and pulmonary complications, which can be detected by point of care ultrasound. The goal is to comprehensively delineate the long term cardiovascular and pulmonary ultrasound findings in recovered COVID-19 patients, identify risks factors for prolonged heart/lung injury, evaluate long term effects of applied treatment, and assess late medication/vaccine side effects in COVID-19 patients.

DETAILED DESCRIPTION:
Aim 1: To examine the long term cardiac involvements of recovered COVID-19 patients at 3, 6, 12 months after being discharged from the hospital or symptom resolution with electrocardiogram (ECG) and echocardiography. 12 lead ECG will be obtained for all patients. Transthoracic echocardiography will be performed using GE Vivid E9 ultrasound system to measure left ventricular (LV) dimensions, LV volumes and LV ejection fraction (EF), wall thickness, LV mass, and LV remodeling index. LV diastolic function will be characterized by maximum velocities of mitral inflow E and A waves, E/A ratio, E/E' ratio (maximum myocardial velocities (E') of the lateral mitral annulus), isovolumetric relaxation time, tricuspid regurgitation velocity, and left atrial volumes. Right-ventricular function will be assessed by tricuspid annular plane systolic excursion (TAPSE), pulmonary acceleration time, and by estimation of systolic pulmonary artery pressure. We will evaluate mitral, aortic, tricuspid and pulmonic valvular stenosis and regurgitation. In addition, speckle tracking echocardiography will be used to detect subclinical impairment of myocardium in patients who have grossly normal LVEF. Lastly, inferior vena cava will be measured to assess patients' volume status.

Aim 2: To evaluate long term pulmonary involvements of recovered COVID-19 patients at 3, 6, 12 months after being discharged from the hospital or symptom resolution with pulse oximetry, bedside spirometry and lung ultrasound. Pulse oximetry, bedside spirometry, and lung ultrasonography (LUS) will be performed for all patients. The pathological LUS features for every zone will be reported as: (1) normal appearance (A lines, < 3 B lines), (2) pathologic B lines (≥3 B lines), (3) confluent B lines, (4) thickening of the pleura with pleural line irregularities (subpleural consolidation < 1 cm), (5) consolidation (≥ 1 cm), (6) pleural effusion. The LUS score, used as a correlate of loss of lung tissue aeration, as well as a normalized LUS score corrected for the number of examined zone, will be calculated in every patient.

Aim 3: To diagnose long term vascular involvements of recovered COVID-19 patients at 3, 6, 12 months after being discharged from the hospital or symptom resolution with vascular ultrasound. A trained physician or sonographer will use high resolution gray-scale imaging, color Doppler ultrasound and spectral analysis with pulse wave Doppler to examine bilateral upper/lower extremity venous and arterial systems and carotid arteries for thrombosis, atheroma, and stenosis.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Consent to participate in this research
* Confirmed SARS-CoV-2 infection by RT-PCR or serological tests.

Exclusion Criteria:

* Refusal to participate in this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Asymptomatic/Mild Group: 50 confirmed COVID-19 patients who showed no or only mild respiratory/GI symptoms; Moderate Group: 50 confirmed COVID-19 patients who were able to maintain oxygen saturation above 92% (or above 90% for patients with chronic lung disease) with up to 4 L/min oxygen via nasal prongs; Severe Group: 50 confirmed COVID-19 patients who had oxygen saturation less than 92% at rest and PaO2/FiO2 between 200 and 300; Critical Group: 50 confirmed COVID-19 patients who had PaO2/FiO2 less than 200 or required mechanical ventilation. Control Group: 50 age and sex-matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
Echocardiographic strain measurements of the left, right heart | Up to 12 months
  strain is a measurement of systolic function of the heart, unit is %. The more negative means better outcome

SECONDARY OUTCOMES:
Lung ultrasound measurements | Up to 12 months
  lung ultrasound scores, B line numbers

OTHER OUTCOMES:
Vascular ultrasound findings | Up to 12 months
  High resolution gray-scale imaging, color Doppler ultrasound and spectral analysis (cm/s) with pulse wave Doppler to examine bilateral upper/lower extremity venous and arterial systems and carotid arteries for thrombosis, atheroma, and stenosis.

CONTACTS AND LOCATIONS:
Overall Officials: Jiapeng Huang, MD, PhD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville Health, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No